CLINICAL TRIAL: NCT03476980
Title: Two Year Developmental Follow-up for Premature Infants Receiving Milking or Delayed Cord Clamping: PREMOD2
Brief Title: Two Year Developmental Follow-up for PREMOD2 Trial (Premature Infants Receiving Milking or Delayed Cord Clamping)
Acronym: PREMOD2FU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sharp HealthCare (Other)
Collaborators: Sharp Mary Birch Hospital for Women & Newborns (Other); Loma Linda University (Other); University of Pittsburgh (Other); Providence Hospital (Other); University of Alabama at Birmingham (Other); University of Alberta (Other); University College Cork (Other); University of Ulm (Other); Christiana Care Health Services (Other); Thrasher Research Fund (Other); Sharp Grossmont Hospital (Other); University of Utah (Other); University of Mississippi Medical Center (Other); PIH Health Good Samaritan Hospital (Unknown); University of California, Irvine (Other); Children's Hospital Medical Center, Cincinnati (Other); Cook County Health (Other Government); St. Louis University (Other); LAC+USC Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: PREMOD2 Follow-Up
Record Dates: First submitted 2018-03-19; First posted 2018-03-26 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-11

CONDITIONS: Neurodevelopmental Abnormality
Keywords: Neurodevelopmental impairment, prematurity; Disability; Umbilical cord milking; Delayed cord clamping
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: Neurodevelopmental assessments will be done at 2 years of corrected age (22-26 months) for subjects who were randomized at birth to receive either delayed cord clamping or umbilical cord milking as part of the PREMOD2 trial. This prospective multi-national randomized controlled trial (RCT) is a two-arm parallel non-inferiority design of two alternative approaches of treatment.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Neurodevelopmental providers will be blinded to the randomization of the toddler during the examination.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Randomized to Umbilical Cord Milking at birth (Active Comparator): Milking the umbilical cord towards the infant at a speed of 20cm/2seconds at birth.
  Interventions: Procedure: Randomized to Umbilical Cord Milking at birth
- Randomized to Delayed Cord Clamping at birth (Active Comparator): Delayed clamping of the umbilical cord at birth.
  Interventions: Procedure: Randomized to Delayed Cord Clamping at birth

INTERVENTIONS:
Procedure: Randomized to Umbilical Cord Milking at birth — The subjects in this group were randomized to UCM X4 at birth. This procedure infuses a placental transfusion of blood by milking the umbilical cord towards the infant at birth.
  Other Names: UCM
  Arms: Randomized to Umbilical Cord Milking at birth
Procedure: Randomized to Delayed Cord Clamping at birth — The subjects in this group were randomized to DCC at birth. At delivery, the obstetrician was instructed to delay clamping of the umbilical cord for 60 seconds.
  Other Names: DCC
  Arms: Randomized to Delayed Cord Clamping at birth

SUMMARY:
An extension of the PREMOD2 trial, the PREMOD2 Follow-Up trial will evaluate the neurodevelopmental outcomes at 22-26 months corrected age of preterm children who received UCM or DCC. This prospective multi-national randomized controlled trial (RCT) is a two-arm parallel non-inferiority design of two alternative approaches of treatment.

DETAILED DESCRIPTION:
The PREMOD2 Follow-up trial will examine the difference in early childhood neurodevelopmental outcomes of subjects enrolled in the PREMOD2 umbilical cord milking (UCM) vs. delayed cord clamping (DCC) trial, using standardized neurologic and developmental assessments at 22-26 months corrected age (CA). The corrected age may be extended out to 42 months CA due to Covid-19 pandemic for undetermined period of time.

ELIGIBILITY:
Inclusion Criteria:

* Children enrolled in the PREMOD2 non-inferiority trial at birth who survive to 2 years corrected age.

Exclusion Criteria:

* Children enrolled in the PREMOD2 non-inferiority trial at birth who did not survive or are lost to follow-up.

Ages: 22 Months to 42 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1200 (Estimated)
Dates: Start 2019-07-06 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Developmental Outcome | 22-26 months corrected gestational age (CGA). All assessments may be extended to 42 months CGA due to Covid-19 pandemic.
  Bayley Scales of Infant Development (BSID), 3rd or 4th Ed. Composite Score (cognitive 55-145, language 45-155, motor 45-155; higher scores are better)

SECONDARY OUTCOMES:
Moderate/Severe Neurodevelopmental Impairment | 22-26 months corrected gestational age
  Defined having at least one of the following: a cognitive score <70, GMFCS greater or equal 2, blindness (vision <20/200), or hearing impairment interfering with the ability to communicate with amplification.
Mild Neurodevelopmental Impairment | 22-26 months corrected gestational age
  Defined having at least one of the following: a cognitive score 70-84, GMFCS =1, unilateral blindness (vision <20/200 in only one eye), or hearing impairment which does not interfere with the ability to communicate.
Gross Motor Function Classification System Scale (GMFCS) | 22-26 months corrected gestational age
  The GMFCS is a validated system used to describe the severity of motor dysfunction. Scale measured from Level 0-5 with Level 0 being normal and Level 5 being the worst score. Measures ability to walk, sit, head control, voluntary movements and postures.
Cerebral Palsy (CP) | 22-26 months corrected gestational age
  Classified as None, Mild, Moderate or Severe based on GMFCS score; No CP = GMFCS Level 0, Mild CP = GMFCS Level 1, Moderate CP = GMFCS Levels 2-3, Severe CP = GMFCS Levels 4-5
Developmental Outcomes assessed by Ages & Stages Questionnaire, 3rd ed. (ASQ-3) five domains: Communication, Gross motor, Fine motor, Problem solving and Personal-social in infants born between 23-32+6 weeks GA who received UCM or DCC. | 22-26 months corrected gestational age
  Each domain is scored from 0 to 60, the higher score is better.
Developmental Outcomes in infants born at 23 -27 and 28-32 weeks GA who received UCM or DCC | 22-26 months corrected gestational age
  BSID Cognitive, Language & Motor composite scores (cognitive 55-145, language 45-155, motor 45-155; higher scores are better) in infants 23-27 weeks GA and 28-32+6 weeks GA.
Developmental Outcomes in infants born at 23 -27 and 28-32 weeks GA who received UCM or DCC | 22-26 months corrected gestational age
  ASQ-3 scores (0 to 60, the higher score is better) in infants 23-27 weeks GA and 28-32+6 weeks GA.
Compare levels of developmental impairment as assessed by BSID-3 or 4 versus the ASQ-3 screening tool. | 22-26 months corrected gestational age
  Mild, moderate or severe impairment
Any grade intraventricular hemorrhage (IVH) in premature newborns 23 - 32+6 weeks GA who received UCM or DCC by mode of delivery (C-Section vs vaginal delivery) | From birth through hospital discharge, up to 6 months corrected gestational age (CGA)
  Any IVH grade from 1 to grade 4, higher grade is worse
Death in premature newborns 23 - 32+6 weeks GA who received UCM or DCC by mode of delivery (C-Section vs vaginal delivery) | From birth through hospital discharge, up to 6 months corrected gestational age (CGA)
  Death
Compare neurodevelopmental outcomes from BSID assessments in newborns 23-32 weeks GA delivered by C-Section with those born by vaginal delivery receiving UCM or DCC. | 22-26 months corrected gestational age
  BSID Cognitive, Language & Motor composite scores (cognitive 55-145, language 45-155, motor 45-155; higher scores are better)
Compare neurodevelopmental outcomes from ASQ assessments in newborns 23-32 weeks GA delivered by C-Section with those born by vaginal delivery receiving UCM or DCC. | 22-26 months corrected gestational age
  ASQ-3 scores (0 to 60, the higher score is better).

OTHER OUTCOMES:
Exploratory, hypothesis-generating | From birth through hospital discharge, up to 6 months corrected gestational age (CGA)
  Any grade IVH, from 1 to 4 (higher is worse)
Exploratory, hypothesis-generating | 4 hours of life +/- 2 hours
  Hemoglobin or Hematocrit at 4 hours of age
Exploratory, hypothesis-generating | In the first 10 minutes of life
  Delivery room interventions received: positive pressure ventilation, continuous positive airway pressure, intubation, chest compressions and medications
Exploratory, hypothesis-generating | In the first 24 hours of life
  Blood pressures in the first 24 hours of life: on admission, 6, 12, 18 and 24 hours of life

CONTACTS AND LOCATIONS:
Overall Officials: Anup Katheria, MD, Principal Investigator — Sharp Mary Birch Hospital for Women & Newborns
Locations (18):
- United States (15):
  - University of Alabama, Birmingham, Alabama
  - Loma Linda Medical Center, Loma Linda, California
  - LAC+USC Medical Center, Los Angeles, California
  - PIH Health Good Samaritan Hospital, Los Angeles, California
  - University of California, Irvine Medical Center, Orange, California
  - Sharp Grossmont Hospital, San Diego, California
  - Sharp Mary Birch Hospital for Women and Newborns, San Diego, California
  - Christiana Care, Newark, Delaware
  - John H. Stroger, Jr. Hospital of Cook County, Chicago, Illinois
  - University of Mississippi Medical Center, Jackson, Mississippi
  - St. Louis University, St Louis, Missouri
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Magee-Womens Hospital, Pittsburgh, Pennsylvania
  - University of Utah, Salt Lake City, Utah
- Governors of University of Alberta, Edmonton, Alberta, Canada
- University of ULM, Ulm, Baden-Wurttemberg, Germany
- Cork University Maternity Hospital, Cork, Ireland

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available per NICHD requirements (National Institute of Child Health and Human Development).
Supporting Information: Study Protocol, SAP
Time Frame: 2 years after primary publication
Access Criteria: An archived dataset with documentation will be made available for additional uses by outside investigators, in collaboration with the study investigators.
URL: http://clinicaltrials.gov

REFERENCES:
- [Background] Katheria A, Garey D, Truong G, Akshoomoff N, Steen J, Maldonado M, Poeltler D, Harbert MJ, Vaucher YE, Finer N. A Randomized Clinical Trial of Umbilical Cord Milking vs Delayed Cord Clamping in Preterm Infants: Neurodevelopmental Outcomes at 22-26 Months of Corrected Age. J Pediatr. 2018 Mar;194:76-80. doi: 10.1016/j.jpeds.2017.10.037. Epub 2017 Dec 12. PMID 29246467
- [Background] Katheria AC, Truong G, Cousins L, Oshiro B, Finer NN. Umbilical Cord Milking Versus Delayed Cord Clamping in Preterm Infants. Pediatrics. 2015 Jul;136(1):61-9. doi: 10.1542/peds.2015-0368. PMID 26122803